CLINICAL TRIAL: NCT04032821
Title: To Evaluate the Effect of Food on the Pharmacokinetic Characteristics of Alkotinib Capsules in Healthy Subjects,A Single Center, Open, Randomized, Single Dose, Two Period, Two Sequence, Crossover Phase I Clinical Trial
Brief Title: To Evaluate the Effect of Food on the Pharmacokinetic Characteristics of Alkotinib Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZGALK003
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-07

CONDITIONS: NSCLC
Keywords: Pharmacokinetics; Alkotinib

STUDY DESIGN:
Intervention Model Description: Each subject was randomly given Alkotinib capsules on an empty stomach or after a meal, and the cleaning period between the two dosages was set as 14 days. The actual dosing time was subject to the original clinical records. After admission to the ward on day -1 (1 day before drug administration), subjects will eat light dinner A 1:1 ratio was randomly assigned to 2 sequences (1=AB, 2=BA). Each subject was subject to two cycles of trials, and the study drug was taken once on an empty stomach or after meal according to the dosing sequence in the randomization table.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkotinib（300mg）First empty stomach, after the meal (Experimental): Alkotinib（300mg），Subjects need to be fasting overnight for at least 10 hours before being warmed to 240 mL on an empty stomach Water service, lunch 4 hours later, dinner 10 hours later.
  Interventions: Drug: Alkotinib（300mg)
- Alkotinib（300mg）After eating first, after fasting (Experimental): Alkotinib（300mg），Subjects need to be fasting for at least 10 hours overnight, starting 30 min before taking the medication A standard meal (800-1000 CAL) can be taken before taking the medicine, and 240 mL warm water can be taken after the meal Lunch hours later, dinner 10 hours later.
  Interventions: Drug: Alkotinib（300mg)

INTERVENTIONS:
Drug: Alkotinib（300mg) — 1. First empty stomach, after the meal.2. After eating first, after fasting.

SUMMARY:
To evaluate the safety and tolerability of food to Alkotinib Capsules in healthy subjects

DETAILED DESCRIPTION:
Alkotinib is an insulin receptor tyrosine kinase inhibitor that selectively inhibits anaplastic lymphoma Kinase and proto-oncogene protein ROS1。Alkotinib is expected to be used in the treatment of ALK positive and ROS1 positive metastatic non-small cell lung Cancer and other cancers include patients with non-small cell lung cancer who are resistant to treatment with the first generation ALK inhibitor, such as kezotinib。

ELIGIBILITY:
Inclusion Criteria:

* sign the informed consent before the clinicaltrial, and fully understand the clinicaltrial content, process and possible adverse event.
* Be able to complete the research according to the clinicaltrial protocol.
* Subjects (including sexual partners) were willing to be screened up to 6 months after the last study drug administration No family planning and voluntary effective contraceptive measures, the specific contraceptive measures see appendix.
* Male and female subjects aged 18 to 55 years (including 18 and 55 years).
* The weight of male subjects should not be less than 50 kg and that of female subjects should not be less than 45 kg. The body of the Body mass index (BMI) = weight (kg)/height 2 (m2), with a BMI of 18~28 kg/m2 range (including critical value).
* Normal or abnormal physical examination and vital signs have n

  * clinical significance.

Exclusion Criteria:

* Smoking more than 5 cigarettes per day during the first 3 months of the study
* Allergic constitution (multiple drug and food allergies).
* A history of drug and/or alcohol abuse (14 units of alcohol per week: 1 unit = beer 285)ML, or liquor 25 mL, or wine 100 mL)
* Blood donation or massive blood loss within 3 months prior to clinical trial screening (> 450ml)
* Any drugs that alter liver enzyme activity were taken 28 days before screening.
* Within 14 days prior to screening，took any prescription, over-the-counter, vitamin products or Herbs.
* Special diet (including dragon fruit, mango, grapefruit, etc.) or drama in 2 weeks，before screening strenuous exercise or other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
* CYP3A inhibitors (e.g., atanavir, talymycin, clarithromycin, etc.), CYP3A inducers (e.g Drugs metabolized by CYP2C8 (such as amodiaquine, silvastatin, etc.) and CYP2C9 metabolism Drugs such as diclofenac, ibuprofen, etc.
* There have been major changes in diet or exercise habits recently.
* Have taken a study drug or participated in a clinical trial of the drug within three months prior to taking the study drug Check.
* A history of dysphagia or any gastrointestinal illness that affects drug absorption, cholecystitis or cholecystectomy In addition to the history;
* Any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or stomach and duodenum Ulcer etc.
* Subjects who could not tolerate standard meals
* Abnormal ecg has clinical significance, or QTc interval >450 ms, or heart rate or pulse < 55 times /Points.
* Any pulmonary disease, including but not limited to interstitial pneumonia, allergic pneumonia, occlusion.Bronchiolitis, pulmonary interstitial fibrosis,interstitial lung disease (ILD), or any pre-existing disease History.
* Female subjects were lactating during the screening period or during the test or had positive serum pregnancy results sex.
* Clinical laboratory examination has clinical significance abnormality, or other clinical findings within 12 months before screening the following diseases (including but not limited to gastrointestinal tract, heart, lung, kidney,Liver, pancreas, nerve, blood, endocrine, tumor, immune, mental or cardiovascular diseases）.
* Screening for viral hepatitis (including hepatitis b and c), AIDS antibody and syphilis spirochete antibody positive.
* Ingested chocolate, any caffeine containing it or the yellow purinate-rich drug 48 hours before taking it.
* Any use of alcohol within 48 hours prior to taking the study drug.
* Positive urine screening or drug use in the past 5 years.
* Subjects considered to have other factors unsuitable for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 120 hours
  Maximum blood concentration
AUC0-t | up to 120 hours
  Area under the plasma concentration - time curve from 0 to the last measurable concentration time point t
AUC0-∞ | up to 6 months
  Area under the concentration - time curve from zero to infinity

SECONDARY OUTCOMES:
Tmax | up to 6 months
  To the maximum blood concentration time
t1/2 | up to 6 months
  Plasma drug half-life
λz | up to 6 months
  14/5000 The rate constant of plasma concentration elimination in terminal phase
CL/F | up to 6 months
  Apparent clearance
VZ/F | up to 6 months
  Apparent volume

CONTACTS AND LOCATIONS:
Overall Officials: yanhua Ding, MD, Study Chair — The First Hospital of Jilin University
Locations (1):
- The first Bethune hospital of jilin university, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial